CLINICAL TRIAL: NCT03233984
Title: Effect of an Environmental Health Education Program on Pregnant Women in Order to Reduce Endocrine Disruptor Exposition : Controled Randomized Trial on Primary Prevention
Brief Title: Effect of an Environmental Health Education Program on Pregnant Women in Order to Reduce Endocrine Disruptor Exposition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREVED
Record Dates: First submitted 2017-06-26; First posted 2017-07-31 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Pregnancy; Endocrine System; Prevention Program
Keywords: bisphenol-A; prevention; endocrine disruptors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Leaflet only (No Intervention): Women will only receive a leaflet about endocrine disruptor at home.
- non immersive program (Active Comparator): In addition of the leaflet, women will sit in the sensibilisation program that will take place in a neutral environment
  Interventions: Behavioral: sensibilisation program "Ma maison, mon environnement santé"
- immersive program (Experimental): In addition of the leaflet, women will si in the sensibilisation program that will take place in an immersive environment
  Interventions: Behavioral: sensibilisation program "Ma maison, mon environnement santé"

INTERVENTIONS:
Behavioral: sensibilisation program "Ma maison, mon environnement santé" — The aim of this program is to spread the awarness about endocrine disruptors through workshops and presentation.
  Arms: immersive program; non immersive program

SUMMARY:
Endocrine disruptors are known as a cancer cause. On pregnant women, it can induce major foetal pathology and impact growth.

Among those molecules, bisphenol-A (BPA) is a plasticizer that can be found on cans and water.

Through a prevention program, the investigators tried to warned pregnant women on endocrine disruptors exposition risks. The goal here is to assess the effectiveness of this program on their fresh products consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18
* Patients living in Poitiers or city around (near the immersive environment)
* Patients on pregnancy and who declared their pregnancy to the authority
* Patients who planned to give birth in Poitiers's hospital, Châtellerault's hospital or Clinique Fief de Grimoire, in Poitiers.
* Patients giving her agreement

Exclusion Criteria:

* Patients planning to move during the study
* Patients under legal protection
* Patients expecting twins
* Patients unable to speak french
* Patients willing to give birth in another hospital than those mentionned before

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
program effectivness | During the pregnancy (second and third trimester)
  Assessing the Effectiveness of the Prevention Program "My Home, My Health Environment" (consists of a series of workshop in the second and third trimesters of pregnancy) in an immersive environment or not, to evaluate the consumption of fresh products according to exposure endocrine disruptors (cans or industrial products).

SECONDARY OUTCOMES:
psychosocial aspects | During the pregnancy (second and third trimester)
  Assess if the program impact any psychosocial aspects, this outcome will be determine with a psychosocial questionary (to do before and after the intervention for compare the results)
Urine concentration | During the pregnancy (second and third trimester)
  Assess if the program has an impact on the urinary endocrine disruptors's concentrations, this outcome will be determine with samples of urine (to do before and after the intervention for comparate the results)
Milk concentration | After the birth of the child (first year)
  Assess the milk endocrine disruptors's concentration difference between women exposed and unexposed to the program
foetal growth | After the birth of the child (first year)
  Study the relation between endocrine disruptors expositions and foetal growth by merging PREVED and EDDS (a previous trial) datas.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Poitiers, Poitiers, France

REFERENCES:
- [Derived] Robalo M, Ayraud-Thevenot S, Migeot V, Gourgues AS, Albouy M, Venisse N. Detection of Endocrine Disruptors in Human Placenta: A Pilot Study on Exposure and Histopathological Findings. Ther Drug Monit. 2025 Dec 9. doi: 10.1097/FTD.0000000000001414. Online ahead of print. PMID 41361687
- [Derived] Ouazzani HE, Rouillon S, Venisse N, Sifer-Riviere L, Dupuis A, Cambien G, Ayraud-Thevenot S, Gourgues AS, Pierre-Eugene P, Pierre F, Rabouan S; DisProSE Group; Migeot V, Albouy-Llaty M. Impact of perinatal environmental health education intervention on exposure to endocrine disruptors during pregnancy-PREVED study: study protocol for a randomized controlled trial. Trials. 2021 Dec 4;22(1):876. doi: 10.1186/s13063-021-05813-5. PMID 34863252